CLINICAL TRIAL: NCT06283641
Title: Multicentre, Single-arm, Non-interventional Regulatory Post- Marketing Surveillance (rPMS) Study to Evaluate the Safety and Effectiveness of Saxenda® for Weight Management in Routine Clinical Practice in Taiwan.
Brief Title: Study to Evaluate the Safety and Effectiveness of Saxenda® for Weight Management in Routine Clinical Practice in Taiwan.
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-7780; U1111-1289-9747 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Saxenda®: Patients with obesity treated with Saxenda® for weight management in routine clinical practice in Taiwan
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Participants will be treated with commercially available Saxenda® according to routine clinical practice at the discretion of the treating physician, following approved label in Taiwan. The decision to initiate treatment with commercially available Saxenda® has been made by the patient and the treating physician before and independently from the decision to participate in this study.
  Other Names: Saxenda®

SUMMARY:
This is a non-interventional study to evaluate the safety and effectiveness of Saxenda® in obese adults and adolescents in Taiwan. The participants will recieve Saxenda® treatment which is a medicine that doctors can already prescribe.

The study will last for about 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female of Taiwanese patients, age above or equal to 12 years who are under Saxenda® treatment or are scheduled to treat with Saxenda® according to approved label in Taiwan based on the clinical judgment of their treating physician.
2. Patients should have baseline (pre-dosing) values, including body height, weight and initial dosage of Saxenda® .
3. The decision to initiate treatment or to have started with commercially available Saxenda® has been made by the patient/Legally Acceptable Representative (LAR) and the physician independently from the decision to join this study.
4. Informed consent obtained before collection of clinical data for this study. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to Saxenda® , the active substance or any of the excipients
2. Previous participation in this study. Participation is defined as having given informed consent in this study.
3. Treatment with any investigational drug within 30 days prior to initiation of Saxenda® treatment.
4. Female patient who is pregnant, breast-feeding, or intends to become pregnant.
5. Patients with a personal or family history of MTC or in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2).
6. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants are patients with obesity treated with Saxenda® for weight management in routine clinical practice in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) by preferred term (PT) | From baseline (week 0) to week 26
  Percent(%)

SECONDARY OUTCOMES:
Number of adverse drug reaction (ADRs) | From baseline (week 0) to week 26
  Number of events
Number of serious adverse events (SAEs) and serious adverse drug reactions (SADRs) | From baseline (week 0) to week 26
  Number of events
Number of unexpected AEs and unexpected ADRs | From baseline (week 0) to week 26
  Number of events
Number of unexpected SAEs and unexpected SADRs | From baseline (week 0) to week 26
  Number of events
Dose and exposure of liraglutide after initiation and reasons if not escalate to liraglutide 3.0 miligram (mg) for maintenance as specified in the product label | From baseline (week 0) to week 26
  Milligram(mg)
Body weight loss Percent (%) (Adult) | From baseline (week 0) to week 13
  Percent (%)
Body weight loss (%) (Adult) | From baseline (week 0) to week 26
  Percent (%)
Body weight loss Kilogram(Kg) (Adult) | From baseline (week 0) to week 13
  Kilogram(Kg)
Body weight loss (kg) (Adult) | From baseline (week 0) to week 26
  Kilogram(Kg)
The proportion of adult subjects losing at least 5% of baseline body weight | At Week 13
  Percent (%)
The proportion of adult subjects losing at least 5% of baseline body weight | At Week 26
  Percent (%)
The proportion of adult subjects losing more than 10% of baseline body weight | At Week 13
  Percent (%)
The proportion of adult subjects losing more than 10% of baseline body weight | At Week 26
  Percent (%)
The proportion of losing at least 5% of baseline body weight from adult subjects whose maintenance dose of 3 mg, 12- week Saxenda® | At Week 26
  Percent (%)
Change in body mass index (BMI) (kg/m^2) (Adolescent) | From baseline (week 0) to week 13
  Kilogram(Kg) divided by meters squared(m2)
Change in body mass index (BMI) (kg/m^2) (Adolescent) | From baseline (week 0) to week 26
  Kilogram(Kg) divided by meters squared(m2)
Change in body mass index (BMI) (%) (Adolescent) | From baseline (week 0) to week 13
  Percent (%)
Change in body mass index (BMI) (%) (Adolescent) | From baseline (week 0) to week 26
  Percent (%)
Change in body mass index standard deviation score (BMI SDS) (Adolescent) | From baseline (week 0) to week 13
  Change in body mass index standard deviation score (BMI SDS)
Change in body mass index standard deviation score (BMI SDS) (Adolescent) | From baseline (week 0) to week 26
  Change in body mass index standard deviation(BMI SDS)
Body weight loss (%) (Adolescent) | From baseline (week 0) to week 13
  Percent (%)
Body weight loss (%) (Adolescent) | From baseline (week 0) to week 26
  Percent (%)
Body weight loss (kg) (Adolescent) | From baseline (week 0) to week 13
  Kilogram(Kg)
Body weight loss (kg) (Adolescent) | From baseline (week 0) to week 26
  Kilogram(Kg)
The proportion of adolescent subjects losing at least 4% of baseline BMI | At Week 13
  Percent(%)
The proportion of adolescent subjects losing at least 4% of baseline BMI | At Week 26
  Percent(%)
The proportion of adolescent subjects losing at least 10% of baseline BMI | At Week 13
  Percent(%)
The proportion of adolescent subjects losing at least 10% of baseline BMI | At Week 26
  Percent(%)
The proportion of losing at least 4% of baseline BMI from adolescent subjects whose maintenance dose of 3 mg or maximum tolerated dose, 12- week Saxenda® | At Week 26
  Percent(%)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (15):
- Taiwan (15):
  - Changhua Christian Hospital_Metabolic Dept., Changhua
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - HsinChu MacKay Memorial Hospital, Hsinchu
  - HsinChu Municipal MacKay Children's Hospital, Hsinchu
  - Ton-Yen General Hospital, Hsinchu County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - TZ Clinic, Pingtung County
  - China Medical University Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - Tungs Taichung MetroHarbor Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital_main, Taipei
  - Genesis Clinic, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com